CLINICAL TRIAL: NCT01873456
Title: Is Multifactorial Nutritional Treatment for Undernutrition in Older Adults in Primary Care Cost-effective?
Acronym: CES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Christian Bitz, Reserarch Director, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CES1
Record Dates: First submitted 2013-05-29; First posted 2013-06-10 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Frail Older Adults
MeSH Terms: interventions — Nutritionists; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifactorial nutritional intervention (Experimental): dietician, resistance type exercise, dysphagia assessment and treatment
  Interventions: Other: multifactorial nutritional intervention
- usual care (No Intervention): usual care

INTERVENTIONS:
Other: multifactorial nutritional intervention
  Other Names: dietician, resitance type exercise, dysphagia assessment and treatment
  Arms: Multifactorial nutritional intervention

SUMMARY:
The hypothesis is that there is a profit potential by implementing a multifactorial nutritional intervention among frail elderly since this will result in an improved nutritional status, functional capacity and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Screening for nutritional risk

Exclusion Criteria:

* terminal condition or do not wish to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Quality of life | up to 6 months
  EuroQol (EQ-5D) is a questionnaire with five questions to be answered in three categories. The five questions deal of movement, self-care, usual activities, pain / discomfort and anxiety / depression and any problems with this

SECONDARY OUTCOMES:
Nutritional status | up to 6 months
  Assessment of weight
Hand grip strength | up to 6 months
  Residents and clients hand grip strength is determined using the dynamometer The dynamometer consists of a narrow handle with two strings as the older must squeezing so hard, they manage three times. The highest value will be used.
Costs | up to 6 months
  Here is used information on additional costs of nutrition efforts, which on the one hand involves all costs associated with the effort, while on the other hand also be seen on the savings that can be attached to the outcome of the effort. Since the purpose is to illustrate the cost-effectiveness, the net profit on the cost side is also compared with the effect of nutritional intervention in terms of improved quality of life, and hence would be able to shed light on efforts from both resource use and a health effect
Activities of Daily Living and cognitive performance | up to 6 months
  Data is collected by Means of the resident assessment instrument
physical strength | up to 6 months
  30 seconds chair stand is used

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Beck, Principal Investigator — University of Copenhagen
Locations (1):
- Home care and nursing homes, Frederiksberg, Denmark

REFERENCES:
- [Background] Beck AM, Keiding H, Christensen AG, Hansen BS, Svendsen SD, et al. (2015) Multidisciplinary Nutritional Support for Page 2 of 7 Undernutrition in Older Adults in Nursing Home and Home-Care is Cost-Effective. SOJ Nur Health Care 1(1): 1-7.
- [Result] Beck AM, Gogsig Christensen A, Stenbaek Hansen B, Damsbo-Svendsen S, Kreinfeldt Skovgaard Moller T, Boll Hansen E, Keiding H. Study protocol: cost-effectiveness of multidisciplinary nutritional support for undernutrition in older adults in nursing home and home-care: cluster randomized controlled trial. Nutr J. 2014 Aug 28;13:86. doi: 10.1186/1475-2891-13-86. PMID 25163483
- [Result] Beck AM, Christensen AG, Hansen BS, Damsbo-Svendsen S, Moller TK. Multidisciplinary nutritional support for undernutrition in nursing home and home-care: A cluster randomized controlled trial. Nutrition. 2016 Feb;32(2):199-205. doi: 10.1016/j.nut.2015.08.009. Epub 2015 Sep 3. PMID 26553461